CLINICAL TRIAL: NCT04891042
Title: The Importance of Isthmocele Development Due to Primary Cesarean Section at The Latent or Active Phase of Labour
Brief Title: Isthmocele Development Due to Primary Cesarean Section at The Latent or Active Phase
Acronym: Isthmocele
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Resul Karakuş, Specialist, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Other Study IDs: 2020/178
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Uterus; Scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Latent Phase of Labour
- Active Phase of Labour

SUMMARY:
The importance of isthmocele development due to primary cesarean section at the latent or active phase of labour

DETAILED DESCRIPTION:
The dates between February 2021 to December 2021 , primiparous (primigravida) and multiparous (multigravida) patients who were hospitalized for delivery between 32 and 41 weeks of gestation and who haven't received cesarean in their previous delivery will be included in the study in Zeynep Kamil Training and Research Hospital Hynecology and Obstetrics Clinic. These patients who will have indication for primary cesarean section will be divided into two groups as latent and active phase according to cervical opening and effacement.During cesarean section , tue uterine lower segment transverse incision will be continuously sutured with 1.0 vicryl( with no interlocking). Also the visceral peritoneum of the vesicle-uterine cavity will be sutured with 2.0 vicryl, This closure technique is to provide hemostasis in the incision. Also additional single interrupted sutures will be recorded(on the each side and /or in the middle of incision).Also If additional surgical interventions such as vessel ligation, uterine artery compression sutures ( such as B-Lynch) will be performed during the surgery, the will be recorded.In this study, If the patients with gestational age below 32, confirmed placenta previa or invasion anomaly and a history of previous cesarean section will not be included.All patient's age, gravid , parity, height, weight, gestational week, smoking history, chronic disease such as hypertension, diabetes mellitus, obstetric history such as oligo-polihidroamnios, abortus imminent,etc previous abdominal surgeries, drug use, use of dinoprost(process) for cervical effacement, cervical Foley catheter use, use of oxytocin, duration of labor, presence of early membrane rupture, time interval from the beginning of rupture membrane, presentation, indication for cesarean section, cervikal dilatation and effacement just before the cesarean section, duration of the operation, use of additional uterotonics during the surgery, additional sutures for hemostasis, presence of atony, additional surgical interventions( uterine artery and hypogastric artery ligation, uterine compression sutures), birth weight, preoperative and post hemogram, hematocrit, white blood cell count, platelet count, blood transfusion if it was given, discharge time, and endometriosis will be recorded. Patients will be called for control examination in the third( 3rd) month after operation. And patients will be asked about clinical findings such as prolonged menstrual bleeding, midsiklus bleeding, dysmenorrhea, pelvic pain. At the same time the presence of isthmuses, the depth and the shape of the istmosel pocket and the myometrial thickness will be measured and recorded with transvaginal ultrasound. Thus, the importance of isthmocele formation on patients who had caeserean section either on latent phase or active phase of labor will be investigated . In addition , other risk factors leading to isthmocele formation will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with the gestational weeks between 32-41 primigravida or multigravida with no history of caesarean section

Exclusion Criteria:

* Gestational age below 32 weeks
* Confirmed Plasenta Previa and/or placental invasion anomalies
* A history Caeserean Section

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Female pregnant patients between 32 and 41 weeks of gestation and who haven't received cesarean in their previous delivery will be included in the study
Study Population: Pregnant Patients at the age of minimum 18 to 45 and with the gestational weeks between 32 to 41, with no history of caesarean section and no confirmed placenta previa and/or invasion anomaly
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-02 (Actual); Study Completion 2021-12-02 (Estimated)

PRIMARY OUTCOMES:
Isthmocele Development | 10 months
  ISTHMOCELE DEVELOPMENT ACCORDİNG TO CERVİCAL DİLATATİON AND EFFACEMENTS

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Maternity and Childrens Training and Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No